CLINICAL TRIAL: NCT02994576
Title: A Single-arm Phase 2 Study of Atezolizumab as Induction Therapy in Stage IB-IIIA Non N2 Resectable and Untreated Non-small Cell Lung Cancer (NSCLC)
Brief Title: Atezolizumab as Induction Therapy in Non-small Cell Lung Cancer
Acronym: PRINCEPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000270-38; 2016/2362 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage IB(≥ 2 cm)-IIIA non N2, resectable and untreated NSCLC (Experimental)
  Interventions: Drug: Atezolizumab
- Comparative cohort (patients receiving standard treatment) (No Intervention)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab, 1200 mg administered I.V. once
  Arms: Stage IB(≥ 2 cm)-IIIA non N2, resectable and untreated NSCLC

SUMMARY:
Based on the efficacy of immunotherapies in advanced disease with a reasonable safety profile/tolerability we could hypothesize that, immunotherapy should work best in the situation of minimal residual disease, Two clinical trials are ongoing to test the role of immunotherapeutic agents in the adjuvant setting: PEARLS trial, a randomized phase III trial with anti-PD1 monoclonal antibody pembrolizumab (MK-3475 or pembrolizumab) versus placebo for patients with early stage NSCLC after resection and completion of standard adjuvant therapy, and the second randomized phase III trial (NCT02273375) will evaluate the efficacy of an anti-PD-L1 (MEDI 4736) for a maximum of 12 months versus placebo as adjuvant therapy in completed resected stage IB-IIIA NSCLC and completed standard ACT.

The role of immunotherapeutic approaches for NSCLC in the neoadjuvant setting is currently unknown. However, based on the survival efficacy of immunotherapeutic strategies in advanced NSCLC where the tumor has not been removed which could produce higher immunogenicity and based on the efficacy of neoadjuvant treatments in NSCLC, we propose to test the safety and efficacy of atezolizumab as neoadjuvant therapy in subjects diagnosed with stage I, II, or IIIA (non N2) NSCLC and who are deemed suitable for surgical resection.

Clinical staging of NSCLC is based on computed tomography (CT) of the chest and upper abdomen, brain CT or magnetic resonance imaging and 18F-FDG PETscan to rule out metastatic disease and assess the potential for curative-intent resection. Adjuvant chemotherapy will be performed according the standard clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the principal study:

* Age ≥ 18 years
* Histologically documented NSCLC
* Clinical Stage IA (≥ 2 cm)-IIIA non N2 NSCLC eligible for surgical resection
* Initial work-up including pet scan and MRI for staging
* Measurable disease, as defined by RECIST v1.1.
* Apt to surgical resection by a lobectomy or bilobectomy procedure
* ECOG performance status of 0 or 1 (appendix 3)
* Adequate hematologic and organ function, defined by the following laboratory results obtained within 14 days prior to registration:

  * White blood cell (WBC) counts > 2.5 x 10^9/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (without granulocyte colony-stimulating factor support within 2 weeks prior to Day 1)
  * Platelet count ≥100 x 10^9/L
  * Hemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase ≤ 2.5 X the upper limit of normal (ULN),
  * Serum bilirubin ≤ 1.5 X ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 X ULN may be enrolled.
  * International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN -This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
  * Creatinine clearance ≥ 60 mL/min on the basis of the Modification of Diet in Renal Disease (MDRD)
  * Serum albumin ≥2.5 g/dL
  * Calcemia ≤ 2.65 mmol/L or Ca ≤10 mg/dL
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days before the registration and must be willing to use two methods of contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for 5 months after last study drug administration. Sexually active males and their female partners must agree to use two methods of accepted and effective contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study.
* Information delivered to the patient and informed consent form signed by the patient
* Ability to comply with the protocol procedures
* Patient affiliated to a social security system or beneficiary of the same

Inclusion criteria for patients included in the comparative cohort (patients receiving standard treatment):

* Age ≥ 18 years
* NSCLC
* Clinical Stage IA (≥2 cm)-IIIA eligible for surgical resection (per the Union Internationale contre le Cancer/American Joint Committee on Cancer staging system, 7th edition; Detterbeck et al. 2009)
* Information delivered to the patient and informed consent form signed by the patient
* Ability to comply with the protocol procedures
* Patient affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

Non-inclusion criteria for the principal study:

Patients who meet any of the following criteria will be excluded from study entry:

* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma for at least five years before registration.
* Prior therapy for lung cancer
* Pregnant and breast feeding women
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary (CHO) cell products or any component of the atezolizumab product
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, Type I diabetes mellitus, vasculitis, or glomerulonephritis (see Appendix 5 for a more comprehensive list of autoimmune diseases). Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* History of HIV infection
* Patients with active hepatitis B (chronic or acute) or hepatitis C Patients with past/resolved HBV infection (defined as the presence of anti-hepatitis B core antibody, IgG anti-HBs + and absence of HbsAg) are eligible. HBV DNA should be obtained in these patients prior to Day 1.

Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.

* Active tuberculosis
* Severe infections within 4 weeks prior to registration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to registration
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Major surgical procedure other than for diagnosis within 28 days prior to registration or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic stem cell or solid organ transplant
* History of any hematological disease not considered in complete remission for at least five years before registration.
* Administration of a live, attenuated vaccine within 4 weeks before registration or anticipation that such a live attenuated vaccine will be required during the study or for 5 months after study drug administration. Influenza vaccination should be given during influenza season only (approximately October to March).

Patients must not receive live, attenuated influenza vaccine (e.g., FluMistâ) within 4 weeks prior to registration or at any time during the study.

* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including but not limited to interferons, interleukin-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior registration
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to registration
* Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the coordinating investigator. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

Non-inclusion criteria for the comparative cohort (patients receiving standard treatment):

* Prior therapy for lung cancer
* Pregnant and breast feeding women
* Active tuberculosis
* Severe infections within 4 weeks prior to registration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to registration
* Prior allogeneic stem cell or solid organ transplant
* History of any hematological disease not considered in complete remission for at least five years before registration.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons, interleukin-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior registration
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to registration
* Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the principal investigator. The use of inhaled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
The rate of patients without major toxicities or morbidities | During the period defined as the start of treatment and 1 month after the surgery (2-month tolerance rate)
  Major toxicities or morbidities: it will include
  a) treatment toxicity leading to a delay of at least 15 days of the surgery, b) grade ≥ 3 toxicity occurring within 2 months after atezolizumab infusion, c) major postoperative morbidity and d) any death related to the experimental treatment and occurring in the period from the day of injection of atezolizumab to the 30 postoperative days. Patients that did not have surgery because of early progression will be considered as having major toxicities or morbidities.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Gustave Roussy, Villejuif, Val De Marne
  - Centre Hospitalier de Chauny, Chauny
  - Centre Marie Lannelongue, Le Plessis-Robinson

IPD SHARING:
Plan to Share IPD: No